**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502a / 71615002

## STATISTICAL ANALYSIS PLAN

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Atopic Dermatitis

Protocol Number: DSXS 1502a Novum Study Number: 71615002

## **Sponsor:**

Taro Pharmaceuticals U.S.A., Inc. 3 Skyline Drive, Hawthorne, NY 10532 USA

## **Contract Research Organization:**

Novum Pharmaceutical Research Services 225 W. Station Square Drive, Suite 200 Pittsburgh, PA 15219

May 19, 2017

Final Version 1.0

Desoximetasone 0.15% Topical Spray

Protocol / Study No. DSXS 1502a / 71615002

## SAP FINAL VERSION APPROVALS

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Atopic Dermatitis

| Written By: Signature: Jianhua Liu, MSc Senior Biostatistician Novum Pharmaceutical Research Services | Date: 06/13/2017 |
|---|---|
| Reviewed By: Signature: Pina D'Angelo, MSc Senior Director, Scientific Affairs (Biostatistics) Novum Pharmaceutical Research Services | Date: 06/13/2017 |
| Approved By: Natalie Signature: Yantovskiy Natalie Yantovskiy Natalie Yantovskiy Senior Director, Clinical Research Taro Pharmaceuticals U.S.A., Inc. | Date: 9 June 2017 |

Desoximetasone 0.15% Topical Spray

Protocol / Study No. DSXS 1502a / 71615002

## **Revision History**

| VERSION | DATE | DESCRIPTION OF REVISIONS | REVISED BY |
|-----------|------------------|--------------------------|-------------|
| Draft 1.0 | January 19, 2017 | New Document | Jianhua Liu |
| Final 1.0 | May 19, 2017 | SAP finalization | Jianhua Liu |

## **Desoximetasone 0.15% Topical Spray**

Protocol / Study No. DSXS 1502a / 71615002

#### List of Abbreviations and Definition of Terms

ADaM Analysis Data Model
AE Adverse Event
BP Blood Pressure
BSA Body Surface Area

C Celsius

CRF Case Report Form

CDISC Clinical Data Interchange Standards Consortium

CRO Contract Research Organization
EASI Eczema Area and Severity Index

F Fahrenheit

FDA Food and Drug Administration

HR Heart Rate Hg Mercury

HPA Hypothalamic Pituitary Adrenal

ICH International Conference on Harmonisation

IGA Investigator's Global Assessment

IND Investigational New Drug

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

ITT Intent-to-Treat

LOCF Last Observation Carried Forward OGD The Office of Generic Drugs

PP Per-Protocol

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAS Statistical Analysis System
SDTM Study Data Tabulation Model
USA United States of America

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502a / 71615002

## TABLE OF CONTENTS

| 1. | INTRODUCTION | 8 |
|---|---|---|
| | OBJECTIVES | |
| | OVERALL STUDY DESIGN | |
| 4. | RANDOMIZATION AND BLINDING | 11 |
| | SAMPLE SIZE | |
| | STUDY ENDPOINTS | |
| 7. | STATISTICAL ANALYSIS METHODS | 12 |
| | 7.1 Baseline Characteristics | 12 |
| | 7.1.1 Subject Disposition | 12 |
| | 7.1.2 Demographic and Other Baseline Characteristics | 12 |
| | 7.1.3 Medical History | 12 |
| | 7.1.4 Concomitant Medications | 13 |
| | 7.1.5 Pregnancy Test | |
| | 7.2 Safety Analysis of Potential HPA Axis Suppression | 13 |
| | 7.3 Safety Analysis | |
| | 7.3.1 Adverse Events | 14 |
| | 7.3.2 Vital Signs | 14 |
| | 7.3.3 Laboratory Evaluations | 14 |
| | 7.3.4 Investigator Global Assessment | 15 |
| | 7.3.5 Eczema Area and Severity Index Score (EASI) | 15 |
| | 7.3.6 Percent BSA Affected | 15 |
| | 7.3.7 Application Site Reaction | 16 |
| | 7.3.8 Pruritus Assessment | 16 |
| | 7.4 Multiple Comparisons | 16 |
| | 7.5 Methods for Handling Missing Data | 16 |
| | 7.6 Interim Analyses | |
| | 7.7 Changes to the Planned Analyses | 16 |
| 8. | TABLE, LISTING AND FIGURE SHELLS | |
| | T16.1.9.1 Summary of Enrolled Patients | 19 |
| | T16.1.9.2 Summary of Protocol Deviations (Safety Population) | 20 |
| | T16.1.9.3 Summary of Demographic Data (Safety Population) | 21 |
| | T16.1.9.4 Summary of Patients Randomized, Included in Safety Analysis of Potential | |
| | HPA Axis Suppression by Study Center | 23 |
| | T16.1.9.5 Summary of Frequency of HPA Axis Suppression at the End of Treatment | |
| | (Day 28) | 24 |
| | T16.1.9.5a Summary of Logistic Regression Analysis Results of HPA Axis | |
| | Suppression at the End of Treatment (Day 28) | 25 |
| | T16.1.9.6 Summary of Percent BSA Affected with Atopic Dermatitis (Safety | |
| | Population) | 26 |
| | T16.1.9.7 Summary of Frequency of Investigator Global Assessment (IGA) (Safety | |
| | Population) | 27 |

| Desoximetasone 0.15% Topical Spray | Protocol / Study No. DSXS 1502a / | 71615002 |
|---|---|---|

| | T16.1.9.8 Summary of Total Score - Eczema Area and Severity Index (EASI) (Safety | |
|---|---|---|
| | Population) | 28 |
| | T16.1.9.9 Overall Summary of Adverse Events (Safety Population) | 29 |
| | T16.1.9.10.1 Summary of Frequency of All Adverse Events by Body System (Safety | |
| | Population) | 30 |
| | T16.1.9.10.2 Summary of Frequency of All Adverse Events in $\geq$ 2% of Patients by | |
| | Body System (Safety Population) | 30 |
| | T16.1.9.11 Summary of Frequency of All Adverse Events by Severity (Safety | |
| | Population) | 31 |
| | T16.1.9.12 Summary of Frequency of All Adverse Events by Relationship (Safety | |
| | Population) | |
| | T16.1.9.13 Summary of Frequency of Serious Adverse Events (Safety Population) | 33 |
| | T16.1.9.14 Summary of Shift Analysis of Clinical Laboratory Assessments | |
| | (Chemistry) from Baseline to Day 28 (Safety Population) | 34 |
| | T16.1.9.15 Summary of Shift Analysis of Clinical Laboratory Assessments | |
| | (Hematology) from Baseline to Day 28 (Safety Population) | 34 |
| | T16.1.9.16 Summary of Frequency of Pruritis Assessment (Safety Population) | 35 |
| | T16.1.9.17 Summary of Application Site Reaction (Safety Population) | 36 |
| | L16.2.1 Listing of Discontinued Patients | 37 |
| | L16.2.2 Listing of Protocol Deviations | 38 |
| | L16.2.3 Patients Excluded from Safety Analysis of Potential HPA Axis Suppression | 39 |
| | L16.2.4.1 Listing of Demographic Data | |
| | L16.2.4.2 Listing of Medical History | 41 |
| | L16.2.4.3 Listing of Concomitant Medication | |
| | L16.2.5.1 Listing of Drug Administration | |
| | L16.2.5.2 Listing of Study Medication Weight | |
| | L16.2.6.1 Listing of Cortisol Response Test Results | |
| | L16.2.6.2 Listing of HPA Axis Suppression Follow-Up | |
| | L16.2.6.3 Listing of Investigator Global Assessment (IGA) | |
| | L16.2.6.4 Listing of Percent BSA Affected with Atopic Dermatitis | |
| | L16.2.6.5 Listing of Eczema Area and Severity Index (EASI) | |
| | L16.2.6.6 Listing of Pruritis Assessment | |
| | L16.2.6.7 Listing of Application Site Reaction | |
| | L16.2.7 Listing of Adverse Events by Cohort | |
| | L16.2.8.1 Listing of Positive Pregnancy Test Results | |
| | L16.2.8.2 Listing of Abnormal Vital Signs | |
| | L16.2.8.3 Listing of Abnormal Physical Examination Results | |
| | L16.2.8.4 Listing of Clinical Hematology Laboratory Results | |
| | L16.2.8.5 Listing of Clinical Chemistry Laboratory Results | |
| ( | D. APPENDICES | |
| | APPENDIX A: Body Surface Area Calculation | |
| | APPENDIX B: Eczema Area and Severity Index Score (EASI) | |
| | APPENDIX C: Investigator Global Assessment (IGA) | |

| ıdy No. DSXS 1502a / 7161500 | P | soximetasone 0.15% Topical Spray |
|------------------------------|-------|------------------------------------|
| 6 | ••••• | APPENDIX D: Cortisol Response Test |

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502a / 71615002

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol DSXS 1502a (Novum Study No. 71615002) Rev. 2 dated 09/06/2016. The SAP provides details on the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

- Final Clinical Study Protocol DSXS 1502a (Novum Study No. 71615002) Rev. 2 dated 09/06/2016
- Case Report Form Version 1.0 for Novum Study No. 71615002

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a patient in this study.

#### 2. OBJECTIVES

- 1. The objective of this study is to evaluate the potential of desoximetasone 0.15% topical spray to suppress HPA axis function in patients with moderate to severe atopic dermatitis.
- 2. The secondary objectives are to evaluate to evaluate the efficacy parameters and adverse event (AE) profiles of desoximetasone 0.15% topical spray administered to patients with moderate to severe atopic dermatitis.

#### 3. OVERALL STUDY DESIGN

This open label, safety study is designed to evaluate the potential for adrenal suppression after treatment with desoximetasone 0.15% topical spray (Taro Pharmaceuticals, U.S.A.), for the treatment of moderate to severe atopic dermatitis.

Approximately 25 to 50 eligible patients with atopic dermatitis that satisfy all eligibility criteria will be enrolled into the study at Visit 1. Patients must be overall in good health. They should have a current diagnosis of moderate to severe atopic dermatitis with IGA score of at least 3 or 4.

Approximately twenty-four (25) to fifty (50) patients stratified by age with a confirmed

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502a / 71615002

diagnosis of moderate to severe atopic dermatitis with:

- **Cohort 1** 10 -20 patients age 12-17 years of age with 10-30% body surface area (BSA) affected
- Cohort 2 5-10 patients age 6-11 years of age with 10-30% body surface area (BSA) affected
- Cohort 3 5-10 patients age 2-5 years of age with 10-30% body surface area (BSA) affected
- **Cohort 4** 5-10 patients 6 months to 1 year of age with 10-30% body surface area (BSA) affected

Cohorts will be enrolled in sequential order. Each cohort will initiate enrollment once the previous cohort has reached the minimum number of patients and a safety analysis has been reviewed. Each cohort will be enrolled based on the availability of patients.

Each cohort will be reviewed for the potential of HPA axis suppression. If at least 50% of patients in a Cohort experience HPA axis suppression, enrollment for that cohort will be stopped and no further cohorts will be initiated. If at least 35% of patients have experienced HPA axis suppression across all cohorts combined during the study, enrollment will be discontinued and no other cohorts will be initiated. Cohort 2 will not begin until safety data has been reviewed for Cohort 1. The same process will be followed for each Cohort until the study is complete. The enrollment in the individual Cohort may not be required if the satisfactory safety data for the same age group was obtained in the study DSXS 1502.

Patients enrolled in the study will apply product twice a day, according to provided instructions, for a total of 28 days.

Patients will attend a total of 3 Clinic Visits as follows:

- Visit 1 (Day 1): Screening/Enrollment
- Visit 2 (Day 14±2): Interim Visit
- Visit 3 (Day 29±2): End of Study or Early Termination

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502a / 71615002

Figure 1 Study Schematic

| | Visit 1 | Visit 2 | Visit 3 | Visit 4 |
|---|---|---|---|---|
| Day | 1 | 14±2 | 29±2 | 42±4 |
| Procedures | Enrollment Before 12 pm | Interim<br>Visit | End of Study/Early Termination Before 12 pm | Telephone<br>Follow-Up<br>Visit |
| Informed Consent | X | | | |
| Medical History and<br>Demographics | X | | | |
| Vital Signs | X | X | X | |
| Pregnancy Test* | X | X | X | |
| Physical Exam | X | | X | |
| % BSA Assessment | X | X | X | |
| IGA Score | X | X | X | |
| EASI Score | X | X | X | |
| Application Site Reactions | X | X | X | |
| Concomitant Medication | X | X | X | |
| Laboratory Evaluations | X | | X | |
| Cortisol Response Test | X | | X | |
| Confirm Inclusion/Exclusion<br>Criteria | X | | | |
| Dispense Sunscreen and<br>Wristband | X | | | |
| Weigh and Dispense Study<br>Drug | X | X | | |
| Collect and Weigh Study Drug | , | X | X | |
| Dispense/Review Patient Diary | X | X | X | |
| Adverse Events | | X | X | X |
| Evaluation of Patient Compliance to the Protocol | | X | X | |

<sup>\*</sup> Pregnancy test will be carried out for females of childbearing potential.

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502a / 71615002

#### 4. RANDOMIZATION AND BLINDING

Patients eligible for enrollment into the study will fall into one of four cohorts:

**Cohort 1** – 10 -20 patients age 12-17 years of age with 10-30% body surface area (BSA) affected

**Cohort 2** – 5-10 patients age 6-11 years of age with 10-30% body surface area (BSA) affected

Cohort 3 – 5-10 patients age 2-5 years of age with 10-30% body surface area (BSA) affected

**Cohort 4** – 5-10 patients 6 months -1 year of age with 10-30% body surface area (BSA) affected

At Visit 1 eligible patients will be enrolled to the study and assigned a patient number.

Cohorts will be enrolled in sequential order. Each cohort will initiate enrollment once the previous cohort has reached the required number of patients and a safety analysis has been reviewed. Each cohort will be enrolled based on the availability of patients.

Each cohort will be reviewed for the potential of HPA axis suppression. If at least 50% of patients in each Cohort experience HPA axis suppression, enrollment for that cohort will be stopped and no further cohorts will be initiated. If at least 35% of patients have experienced HPA axis suppression across cohorts combined during the study, enrollment will be discontinued and no other cohorts will be initiated. Cohort 2 will not begin until safety data has been reviewed for Cohort 1. The same process will be followed for each Cohort until the study is complete.

The enrollment in the individual Cohort may not be required if the satisfactory safety data for the same age group was obtained in the study DSXS 1502.

#### 5. SAMPLE SIZE

The sample size of 35 patients, stratified by age and % BSA, was determined to be sufficient.

#### 6. STUDY ENDPOINTS

#### **Primary Outcome Measures:**

Hypothalamic Pituitary Adrenal (HPA) Axis Response to Cosyntropin demonstrating the absence or presence of adrenal suppression at the end of treatment

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502a / 71615002

#### **Secondary Outcome Measures:**

Hypothalamic Pituitary Adrenal (HPA) Axis Response to Cosyntropin demonstrating the presence of adrenal suppression at the end of treatment with % BSA as a covariate.

#### 7. STATISTICAL ANALYSIS METHODS

If not otherwise specified, statistical significance is defined as p<0.05 and is two-tailed. Data will be summarized with respect to demographic and baseline characteristics and safety variables.

For categorical variables, the number and percent of each category within a parameter will be calculated for non-missing data. For continuous variables, statistics will include n, mean, standard deviation, median, minimum and maximum values.

All statistical analyses will be conducted using SAS<sup>®</sup>, Version 9.4 or higher. Datasets will be prepared using headings from Clinical Data Interchange Consortium (CDISC) Study Data Tabulation Model (SDTM) implementation for human clinical trials and ADaM (Analysis Dataset Model).

#### 7.1 Baseline Characteristics

#### 7.1.1 Subject Disposition

The subject accountability and disposition information will be summarized by study cohort. The number of subjects enrolled, treated with study medication will be tabulated by study cohort. In addition, completion status and primary reason for withdrawal will be summarized by study cohort.

## 7.1.2 Demographic and Other Baseline Characteristics

The cohorts will be compared for basic demographics (age, gender, ethnicity and race), baseline IGA, baseline EASI and baseline total BSA.

Summary tables by cohort will be presented. Continuous variables will be summarized using descriptive statistics (n, mean, standard deviation, median, minimum, maximum). Categorical variables will be summarized using frequencies and percentage.

Baseline comparability of the four cohorts will be presented using Chi-square test for the categorical variables, and Analysis of Variance for the continuous variables.

All data will be listed by cohort and patient.

#### 7.1.3 Medical History

At Visit 1, patients will be questioned about medical history, including acute and chronic

## **Desoximetasone 0.15% Topical Spray**

Protocol / Study No. DSXS 1502a / 71615002

medical history and medical history relevant to their atopic dermatitis.

Medical history data will be listed by cohort and patient.

#### 7.1.4 Concomitant Medications

At Visits 1-3, patients will be questioned about current and concomitant medication over the past 12 weeks.

All prior and concomitant medications taken since screening until the end of the study will be listed by cohort and patient.

#### 7.1.5 Pregnancy Test

Urine pregnancy tests on women of child-bearing potential will be performed at Visits 1, 2, and 3.

Positive pregnancy test results will be listed by cohort and patient.

## 7.2 Safety Analysis of Potential HPA Axis Suppression

Dosing will be twice a day for 28 days excluding the doses prior to the Cortisol Response Test (54 applications). All patients who are enrolled, use at least 42 doses of the study drug and have data from a post-treatment cortisol response test will be included in the analysis. Patients who have not used 42 doses of the study drug will be excluded from the primary analysis of HPA axis suppression.

The primary analysis of interest is the proportion of patients in each group who are considered to have demonstrated possible HPA axis suppression following treatment with the study medication. As a secondary analysis of the data a logistic regression of the proportion of patients in the study with HPA axis suppression may be performed with %BSA affected as a covariate. This will depend on the distribution of the %BSA data collected.

The study will be enrolled by Cohort starting with Cohort 1 and each cohort will be reviewed for the potential of HPA axis suppression. If at least 50% of patients in Cohort 1 experience HPA axis suppression once the minimum number of patients has been enrolled and completed the cohort, enrollment for that cohort will be stopped and no further cohorts will be initiated. If at least 35% of patients have experienced HPA axis suppression across cohorts combined during the study, enrollment will be discontinued and no other cohorts will be initiated. Cohort 2 will not begin until safety data has been reviewed for Cohort 1. The same process will be followed for each Cohort until the study is complete.

For all patients the actual amount of desoximetasone (mg) applied during the study will be

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502a / 71615002

calculated from recorded bottle weights and presented.

## 7.3 Safety Analysis

Safety analysis will be conducted on all patients who applied at least one dose of study drug.

#### 7.3.1 Adverse Events

All the adverse events (AEs) reported throughout the study will be coded and classified according to the MedDRA (Medical Dictionary for Regulatory Activities) coding dictionary (Version 19 or higher). Each adverse event is to be evaluated for date of start and end, seriousness, severity, causal relationship with the study drugs, action taken and outcome.

A summary table of the number and percent of patients with AEs by system organ class, preferred term, and cohort will be presented. Each patient will be counted only once within each preferred term.

A frequency summary table of the number of AEs by system organ class, preferred term, severity, and cohort will be presented. Severity will be classified as "Mild", "Moderate", or "Severe".

Similarly, a frequency summary table of the number of AEs by system organ class, preferred term, and relationship to a study drug, and cohort will be presented. Relationship to a study drug will be classified as "Not Related" or "Related" where "Related" includes "Possible", "Probable", or "Definite".

Should sufficient data exist, adverse event frequencies will be compared between cohorts using Fisher's exact test.

All AEs will be listed by cohort and patient.

#### 7.3.2 Vital Signs

The patient's vital signs will be recorded (heart rate, blood pressure, temperature and respiration rate) at Visit 1, 2, and 3.

Abnormal vital signs will be listed by cohort and patient.

#### 7.3.3 Laboratory Evaluations

At Visit 1 and Visit 3 a blood sample will be collected for hematology and clinical chemistry testing. The testing panel should include as a minimum the following tests:

#### Hematology

## **Desoximetasone 0.15% Topical Spray**

Protocol / Study No. DSXS 1502a / 71615002

- Hematocrit
- White blood cell count
- Platelets
- Hemoglobin
- Red blood cell count
- Differential white cell count

#### Chemistry

- Alkaline phosphatase
- Total bilirubin
- Alanine transaminase
- Creatinine
- Aspartate transaminase
- Glucose
- Blood urea nitrogen

Shift analysis using the categories; below, above and within the laboratory normal range will be performed to identify any specific laboratory parameter that shows a trend toward potentially clinically significant changes.

All data will be listed by cohort and patient.

#### 7.3.4 Investigator Global Assessment

At each visit the Investigator will perform an Investigator Global Assessment (IGA).

Investigator Global Assessment will be summarized using frequency and percentage by cohort and visit.

Investigator Global Assessment will also be listed by cohort and patient.

## 7.3.5 Eczema Area and Severity Index Score (EASI)

Eczema Area and Severity Index Score will be assessed at each visit.

EASI will be summarized using frequency and percentage by cohort and visit. EASI will also be listed by cohort and patient.

#### 7.3.6 Percent BSA Affected

The % BSA recorded at Visit 1, 2, and 3 will be summarized descriptively by cohort and visit.

All data will be listed by cohort and patient.

## **Desoximetasone 0.15% Topical Spray**

Protocol / Study No. DSXS 1502a / 71615002

#### 7.3.7 Application Site Reaction

A frequency summary table comparing application site reaction for each cohort will be presented by visit.

All data will be listed by cohort and patient.

#### 7.3.8 Pruritus Assessment

A frequency summary table comparing the severity of pruritus for each cohort will be presented by visit.

All data will be listed by cohort and patient.

#### 7.4 Multiple Comparisons

No multiple comparison adjustment will be made in this study.

## 7.5 Methods for Handling Missing Data

For demographic and baseline characteristics, each variable will be analyzed using all available data. Patients with missing data will be excluded only from analyses for which data are not available.

#### 7.6 Interim Analyses

There is no interim analysis planned in this study.

#### 7.7 Changes to the Planned Analyses

Protocol Section 10.1.3 states as a secondary analysis of the data a logistic regression of the proportion of patients in the study with HPA axis suppression will be performed with %BSA affected as a covariate. The following will be applied during the analyses.

As a secondary analysis of the data a logistic regression of the proportion of patients in the study with HPA axis suppression may be performed with %BSA affected as a covariate. This will depend on the distribution of the %BSA data collected.

## 8. TABLE, LISTING AND FIGURE SHELLS

The following shells are provided in order to provide a framework for the display of data from this study. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables, Listings and Figures that will be included in the final

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502a / 71615002

clinical study report. Tables, Listings and Figures are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. All descriptive and inferential statistical analyses will be performed using SAS® statistical software Version 9.4 or higher, unless otherwise noted.

TABLE, LISTING AND FIGURE SHELLS

**T16.1.9.1 Summary of Enrolled Patients** 

| Patients | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|-------------------|----------|----------|----------|----------|-------|
| Screened | | | | | XXX |
| Randomized | XXX | XXX | XXX | xxx | xxx |
| Completed Study | XXX | xxx | XXX | xxx | XXX |
| Terminated Early | xxx | xxx | xxx | XXX | xxx |
| Adverse Event | xxx | xxx | XXX | xxx | xxx |
| Enrolled in error | xxx | xxx | XXX | xxx | xxx |
| Lack of efficacy | XXX | XXX | XXX | xxx | xxx |
| Lost to follow-up | XXX | xxx | xxx | xxx | XXX |
| etc. | | | | | |
| Other | xxx | xxx | xxx | xxx | xxx |

T16.1.9.2 Summary of Protocol Deviations (Safety Population)

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| Total Patients with Protocol Deviations | XXX | XXX | xxx | XXX | XXX |
| Total Deviations | xxx | xxx | xxx | xxx | xxx |
| Enrolled in Error | xxx | xxx | xxx | xxx | xxx |
| Lost to Follow-up | xxx | XXX | xxx | XXX | xxx |
| Missed Visit | xxx | XXX | XXX | xxx | XXX |
| Non-compliance with study drug | XXX | XXX | xxx | XXX | xxx |
| Outside Visit Window | xxx | XXX | xxx | XXX | xxx |
| Restricted Medication Use | xxx | XXX | xxx | XXX | xxx |
| etc | | | | | |
| Other | xxx | xxx | xxx | xxx | XXX |

Page 1 of N

05/19/2017

T16.1.9.3 Summary of Demographic Data (Safety Population)

| | | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total | <b>3</b> 5. • |
|---|---|---|---|---|---|---|---|
| | | N=xx | N=xx | N=xx | N=xx | N=xx | P-value |
| Age (years) | n | XX | XX | XX | XX | xx | x.xxxx |
| | Mean $\pm$ SD | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | |
| | Median | xx.x | XX.X | xx.x | xx.x | xx.x | |
| | Range | xx-xx | xx-xx | xx-xx | xx-xx | xx-xx | |
| Age Groups | <=1 | - | - | - | xx (xx.x%) | - | |
| | 2 - 5 | | - | xx (xx.x%) | - | - | |
| | 6-11 | - | xx (xx.x%) | - | - | - | |
| | 12 - 17 | xx (xx.x%) | - | - | - | - | - |
| | 18 - 40 | - | - | - | - | - | |
| | 41 - 64 | - | - | - | - | · <b>-</b> | |
| | 65 - 75 | - | - | - | - | - | |
| | > 75 | - | - | - | - | - | |
| Race | American Indian or Alaska Native | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | x.xxxx |
| | Asian | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Black/African American | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Native Hawaiian or other Pacific Islander | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | White | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Ethnicity | Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | x.xxxx |
| | Not Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

N= number of patients in the cohort; n= number of patients with data available; % is based on N

Created on: ddmmmyy hh:mm

T16.1.9.3 Summary of Demographic Data (Safety Population)

| | | Cohort 1<br>N=xx | Cohort 2<br>N=xx | Cohort 3 N=xx | Cohort 4<br>N=xx | Total<br>N=xx | P-value |
|---|---|---|---|---|---|---|---|
| Baseline Total BSA | n | XX | XX | XX | XX | xx | x.xxxx |
| | $Mean \pm SD$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | |
| | Median | XX.X | xx.x | xx.x | XX.X | XX.X | |
| | Range | xx-xx | xx-xx | xx-xx | xx-xx | xx-xx | |
| Baseline IGA | Clear | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | x.xxxx |
| | Almost Clear | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| EASI | n | xx | xx | XX | xx | xx | x.xxxx |
| | $\text{Mean} \pm \text{SD}$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | |
| | Median | xx.x | xx.x | xx.x | xx.x | XX.X | |
| | Range | xx-xx | xx-xx | xx-xx | xx-xx | xx-xx | |

N= number of patients in the cohort; n= number of patients with data available; % is based on N

Created on: ddmmmyy hh:mm

T16.1.9.4 Summary of Patients Randomized, Included in Safety Analysis of Potential HPA Axis Suppression by Study Center

| Site | | Total | | | Cohort 1 Cohor | | hort 2 | Cohort 3 | | | Cohort 4 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| No. | PI Name | Rando-<br>mized | Included | Rando-<br>mized | Included | Rando-<br>mized | Included | Rando-<br>mized | Included | Rando-<br>mized | Included |
| All | • | xx | xx(xx.x%) | XX | xx(xx.x%) | xx | xx(xx.x%) | XX | xx(xx.x%) | XX | xx(xx.x%) |
| xx | xxxx | xx | xx (xx.x%) | xx | xx(xx.x%) | xx | xx(xx.x%) | xx | xx(xx.x%) | xx | xx(xx.x%) |
| XX | XXXX | XX | xx(xx.x%) | XX | xx(xx.x%) | XX | xx(xx.x%) | XX | xx(xx.x%) | xx | xx(xx.x%) |

T16.1.9.5 Summary of Frequency of HPA Axis Suppression at the End of Treatment (Day 28)

| HPA Axis<br>Suppression | All<br>N=xx | Cohort 1<br>N=xx | Cohort 2<br>N=xx | Cohort 3<br>N=xx | Cohort 4<br>N=xx |
|---|---|---|---|---|---|
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

T16.1.9.5a Summary of Logistic Regression Analysis Results of HPA Axis Suppression at the End of Treatment (Day 28)

| | Odds Ratio | 95% Wald Confidence Limits | Wald<br>Chi-Square | P-value |
|---|---|---|---|---|
| Cohort 1 vs. Cohort 2 | x.xxxx | x.xxxx, x.xxxx | X.XXXX | x.xxxx |
| Cohort 1 vs. Cohort 3 | x.xxxx | x.xxxx, x.xxxx | x.xxxx | x.xxxx |
| Cohort 1 vs. Cohort 4 | x.xxxx | x.xxxx, x.xxxx | x.xxxx | x.xxxx |
| Cohort 2 vs. Cohort 3 | x.xxxx | x.xxxx, x.xxxx | x.xxxx | x.xxxx |
| Cohort 2 vs. Cohort 4 | x.xxxx | x.xxxx, x.xxxx | x.xxxx | x.xxxx |
| Cohort 3 vs. Cohort 4 | x.xxxx | x.xxxx, x.xxxx | x.xxxx | x.xxxx |
| Baseline % BSA affected | x.xxxx | x.xxxx, x.xxxx | x.xxxx | x.xxxx |

T16.1.9.6 Summary of Percent BSA Affected with Atopic Dermatitis (Safety Population)

| | | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 |
|---|---|---|---|---|---|
| Visit | Statistic | (N = xx) | (N = xx) | (N = xx) | (N = xx) |
| 1 | n | xx | xx | xx | xx |
| | $Mean \pm SD$ | $xxx.x \pm xxx.x$ | $xxx.x \pm xxx.x$ | $xxx.x \pm x xx.x$ | $xxx.x \pm xxx.x$ |
| | Median | xxx.x | xxx.x | xxx.x | xxx.x |
| | Range | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x | XXX.X - XXX.X |
| 2 | | | | | |
| 3 | | | | | |

T16.1.9.7 Summary of Frequency of Investigator Global Assessment (IGA) (Safety Population)

| Visit | Score | Cohort 1 $(N = xx)$ | Cohort 2 $(N = xx)$ | Cohort 3 $(N = xx)$ | Cohort 4 $(N = xx)$ |
|---|---|---|---|---|---|
| | 0 (Clear) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 1 (Almost Clear) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 2 (Mild Disease) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 3 (Moderate Disease) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 4 (Severe Disease) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | 0 (Clear) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 1 (Almost Clear) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 2 (Mild Disease) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 3 (Moderate<br>Disease) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 4 (Severe Disease) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

3

Created on: ddmmmyy hh:mm

T16.1.9.8 Summary of Total Score - Eczema Area and Severity Index (EASI) (Safety Population)

| Visit | Statistic | Cohort 1 $(N = xx)$ | Cohort 2 $(N = xx)$ | Cohort 3 $(N = xx)$ | Cohort 4 $(N = xx)$ |
|---|---|---|---|---|---|
| 1 | n | xx | xx | xx | XX |
| | $Mean \pm SD$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ |
| | Median | xxx.x | xxx.x | xxx.x | xxx.x |
| | Range | xxx - xxx | xxx - xxx | xxx - xxx | xxx - xxx |
| 2 | | | | | |
| 3 | | | | | |

T16.1.9.9 Overall Summary of Adverse Events (Safety Population)

| Description of the second of t | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| Description | N=xx | N=xx | N=xx | N=xx | N=xx |
| Patients Randomized | XXX | xxx | xxx | xxx | XXX |
| Patients with at least one AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued study drug due to above AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| AEs reported | xxx | xxx | xxx | xxx | xxx |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serious AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Related = Possible, Probable, Definite

Created on: ddmmmyy hh:mm

T16.1.9.10.1 Summary of Frequency of All Adverse Events by Body System (Safety Population)

| Body System | MedDRA Term | Cohort | Events | Patients | · Fisher's p-value |
|---|---|---|---|---|---|
| Patients with at least one AE | Total | Cohort 1 (N=xx) | XX | xx (xx.x%) | x.xxxx |
| | | Cohort 2 (N=xx) | XX | xx (xx.x%) | |
| | | Cohort 3 (N=xx) | XX | xx (xx.x%) | |
| | | Cohort 4 (N=xx) | XX | xx (xx.x%) | |
| Ear and labyrinth disorders | Ear pain | Cohort 1 (N=xx) | XX | xx (xx.x%) | x.xxxx |
| | | Cohort 2 (N=xx) | XX | xx (xx.x%) | |
| | | Cohort 3 (N=xx) | XX | xx (xx.x%) | |
| | | Cohort 4 (N=xx) | XX | xx (xx.x%) | |

N = Total number of patient in each cohort; Percentage is based on total number of patients.

T16.1.9.10.2 Summary of Frequency of All Adverse Events in ≥ 2% of Patients by Body System (Safety Population)

T16.1.9.11 Summary of Frequency of All Adverse Events by Severity (Safety Population)

| Body System | MedDRA Term | Cohort | Mild | Moderate | Severe |
|---|---|---|---|---|---|
| Patients with at least one AE | Total | Cohort 1 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 2 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 3 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 4 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth disorders | Ear pain | Cohort 1 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 2 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 3 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 4 (N=xx) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

N = Total number of events in each cohort; Percentage is based on total number of events.

Created on: ddmmmyy hh:mm

T16.1.9.12 Summary of Frequency of All Adverse Events by Relationship (Safety Population)

| <b>Body System</b> | MedDRA Term | Cohort | Related | Not Related |
|---|---|---|---|---|
| Patients with at least one AE | Total | Cohort 1 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 2 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 3 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 4 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth disorders | Ear pain | Cohort 1 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 2 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| • | | Cohort 3 (N=xx) | xx (xx.x%) | xx (xx.x%) |
| | | Cohort 4 (N=xx) | xx (xx.x%) | xx (xx.x%) |

N = Total number of events in each cohort; Percentage is based on total number of events. Related = Possible, Probable, Definite

Created on: ddmmmyy hh:mm

T16.1.9.13 Summary of Frequency of Serious Adverse Events (Safety Population)

| Body System | MedDRA | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 |
|---|---|---|---|---|---|
| | Term | N=xx | N=xx | N=xx | N=xx |
| Injury, poisoning and procedural complications | Alcohol poisoning | xx | xx | xx | xx |

T16.1.9.14 Summary of Shift Analysis of Clinical Laboratory Assessments (Chemistry) from Baseline to Day 28 (Safety Population)

## Alanine Aminotransferase (U/L)

| | | Cohort 1<br>(N=xx) | | | Cohort 2<br>(N=xx) | | | Cohort 3<br>(N=xx) | | - | Cohort 4<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Baseline-><br>Endpoint | Low | Normal | High | Low | Normal | High | Low | Normal | High | Low | Normal | High |
| Low | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| Normal | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |
| High | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) | (xx.x%) |

Table will continue for other lab parameters.

Similar table will be created for T16.1.9.18.

T16.1.9.15 Summary of Shift Analysis of Clinical Laboratory Assessments (Hematology) from Baseline to Day 28 (Safety Population)

T16.1.9.16 Summary of Frequency of Pruritis Assessment (Safety Population)

| Visit | Score | Cohort 1 $(N = xx)$ | Cohort 2 $(N = xx)$ | Cohort 3 $(N = xx)$ | Cohort 4 $(N = xx)$ |
|---|---|---|---|---|---|
| 1 | None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

3

Created on: ddmmmyy hh:mm

T16.1.9.17 Summary of Application Site Reaction (Safety Population)

| Sign / Symptom | Visit | Statistic | Cohort 1 $(N = xx)$ | Cohort 2 $(N = xx)$ | Cohort 3 $(N = xx)$ | Cohort 4 $(N = xx)$ |
|---|---|---|---|---|---|---|
| Burning | 1 | Absent | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | 2 | | | | | |
| | 3 | | | | | |
| Erosion | | | | | | |
| Erosion | | | | | | |
| Edema | | | | | | |
| Pain | | | | | | |
| Itching | | | | | | |
| Dryness | | | | | | |
L16.2.1 Listing of Discontinued Patients

| Cohort | Patient<br>Number | Discontinuation<br>Reason |
|----------|-------------------|---------------------------|
| Cohort 1 | xx-xxxx | Withdrawal by Subject |
| | xx-xxxx | Lost to Follow-up |
| Cohort 2 | | |
| Cohort 3 | | |
| Cohort 4 | | |

## L16.2.2 Listing of Protocol Deviations

| Cohort | Patient<br>Number | <b>Event Description</b> |
|----------------------|-------------------|--------------------------------|
| Cohort 1 | xx-xxxx | Outside Visit Window (Visit 3) |
| Cohort 2<br>Cohort 3 | | |
| Cohort 4 | | |

Created on: ddmmmyy hh:mm

L16.2.3 Patients Excluded from Safety Analysis of Potential HPA Axis Suppression

| Cohort | Patient<br>Number | Exclusion Reason |
|---|---|---|
| Cohort 1 | XX-XXXX | Patient has not used 42 doses of the study drug |
| | | • • |
| Cohort 2 | | |
| Cohort 3 | | |
| Cohort 4 | | |

## L16.2.4.1 Listing of Demographic Data

| Cohort | Patient<br>Number | Age | Gender | Ethnicity | Race |
|---|---|---|---|---|---|
| Cohort 1 | XX-XXXX | 11 | Female | Not Hispanic or Latino | Black or African American |
| 0.10 | | | | | |
| Cohort 2 | | | | | |
| Cohort 3 | | | | | |
| Cohort 4 | | | | | |

Created on: ddmmmyy hh:mm

Page 1 of N

05/19/2017

## L16.2.4.2 Listing of Medical History

| Cohort | Patient<br>Number | System | Diagnosis or<br>Surgical<br>Procedure | Start Date | End Date | Ongoing |
|---|---|---|---|---|---|---|
| Cohort 1 | xx-xxxx | Gynecologic | Menopause | yyyy-mm-dd | yyyy-mm-dd | |
| ~ . | | | | | | |
| Cohort 2 | | | | | | |
| Cohort 3<br>Cohort 4 | | | | | | |
| Conort 1 | | | | | | |

Created on: ddmmmyy hh:mm

# L16.2.4.3 Listing of Concomitant Medication

| Cohort | Patient<br>Number | Treatment<br>Area | Medication | Dosage | Frequency | Route | Start/End<br>Date | Indication |
|---|---|---|---|---|---|---|---|---|
| Cohort 1 | xx-xxxx | No | Lisinopril | 20 MG | QD | PO | yyyy-mm-dd /<br>yyyy-mm-dd | Hypertension |
| Cohort 2<br>Cohort 3<br>Cohort 4 | | | | | | | | |

Created on: ddmmmyy hh:mm

## L16.2.5.1 Listing of Drug Administration

| Cohort | Patient | Date of | Date of | Total | Compliance |
|----------|---------|------------|------------|---------------|------------|
| | Number | First Dose | Last Dose | Doses Applied | (%) |
| Cohort 1 | XXXX | yyyy-mm-dd | yyyy-mm-dd | XX | xx.x |

Cohort 2

Cohort 3

Cohort 4

#### Note to programmer:

Compliance = [Total number of applications] / [Planned number of applications] \* 100%, where Planned number of applications is determined as follows:

for subjects who completed the study successfully: 56 applications (28 days of twice daily dosing);

for subjects who discontinued early: the minimum between 56 and [(Date of Discontinuation – Date of First Application)].

Created on: ddmmmyy hh:mm

L16.2.5.2 Listing of Study Medication Weight

| | | Bott | le 1 | Bottle | 2 | Total |
|---|---|---|---|---|---|---|
| Cohort | Patient<br>Number | Date<br>Dispensed | Weight<br>Dispensed<br>(g) | Date<br>Collected | Weight<br>Collected<br>(g) | Amount<br>Applied<br>(g) |
| Cohort 1 | xxxx | yyyy-mm-dd | XX | yyyy-mm-dd | xx | XXX |

Cohort 2

Cohort 3

Cohort 4

Created on: ddmmmyy hh:mm

## L16.2.6.1 Listing of Cortisol Response Test Results

#### Cohort 1

| Patient<br>Number | Visit | Was a Cortisol<br>Response Test<br>conducted? | | Basal<br>Sample<br>Draw Time | Injection<br>Time | Post-<br>Injection<br>Draw<br>Time | Basal<br>Cortisol<br>Concentration<br>Level<br>(mcg/100ml) | Post Injection<br>Cortisol<br>Concentration<br>Level<br>(mcg/100ml) | | Have<br>HPA Axis<br>Suppression<br>? |
|---|---|---|---|---|---|---|---|---|---|---|
| xx-xxxx | 1 | Yes | yyyy-mm-dd | hh:mm | hh:mm | hh:mm | XXX | XXX | No | |
| | 3 | Yes | yyyy-mm-dd | hh:mm | hh:mm | hh:mm | XXX | XXX | | No |

Table will continue for other cohorts.

Created on: ddmmmyy hh:mm

## L16.2.6.2 Listing of HPA Axis Suppression Follow-Up

| | | | Cohort 1 | | | | |
|---|---|---|---|---|---|---|---|
| Patient<br>Number | Is The Patient Showing Signs<br>Or Symptoms Of HPA Axis<br>Suppression?/<br>Was a Cortisol Response<br>Test Conducted? | Follow-Up<br>Test | Date/<br>Basal Sample Draw Time/<br>Injection Time/<br>Post-Injection Draw Time | Basal<br>Cortisol<br>Concentration<br>Level<br>(mcg/100ml) | Post Injection<br>Cortisol<br>Concentration<br>Level<br>(mcg/100ml) | Still Show Signs of HPA Axis Suppression? | Was the Patient Referred to an Endocrinologist |
| XX-XXXX | Yes/ Yes | Test 1 | yyyy-mm-dd / hh:mm /<br>hh:mm/ hh:mm | XXX | XXX | No | No |

Table will continue for other cohorts.

Created on: ddmmmyy hh:mm

L16.2.6.3 Listing of Investigator Global Assessment (IGA)

| Cohort | Patient<br>Number | Visit 1 | Visit 2 | Visit 3 / Early<br>Termination |
|---|---|---|---|---|
| Cohort 1 | xx-xxxx | 0 | 0 | 0 |
| Cohort 2 | | | | |
| Cohort 3<br>Cohort 4 | | | | |

# L16.2.6.4 Listing of Percent BSA Affected with Atopic Dermatitis

| Cohort 1 xx-xxxx xxx xxx xxx xxx xxx xxx x.xx Cohort 2 Cohort 3 Cohort 4 | Cohort | Patient<br>Number | Visit 1 | Visit 2 | Visit 4 / Early<br>Termination | Baseline Total<br>BSA (m^2) |
|---|---|---|---|---|---|---|
| Cohort 3 | Cohort 1 | xx-xxxx | XXX | XXX | XXX | x.xx |
| Cohort 3 | | | | | | |
| | Cohort 2 | | | | | |
| Cohort 4 | | | | | | |
| | Cohort 4 | | | | | |

Created on: ddmmmyy hh:mm

L16.2.6.5 Listing of Eczema Area and Severity Index (EASI)

| Cohort | Patient<br>Number | Visit | Location | Erythema | Induration,<br>Papulation,<br>Edema | Lichenification | Excoriation | Total<br>Grade | Total<br>EASI<br>Score |
|---|---|---|---|---|---|---|---|---|---|
| Cohort 1 | xx-xxxx | 1 | Head/Neck | 0 | 0 | 0 | 0 | 0 | XXXX |
| | | | Upper Limbs | 0 | 0 | 0 | 0 | 0 | |
| | | | Trunk | 1 | 1 | 1 | 1 | 4 | |
| | | | Lower Limbs | 0 | 0 | 0 | 0 | 0 | |
| | | 2 3 | | | | | | | |
| Cohort 2<br>Cohort 3<br>Cohort 4 | | | | | | | | | |

## L16.2.6.6 Listing of Pruritis Assessment

| Cohort | Patient<br>Number | Visit 1 | Visit 2 | Visit 3/Early<br>Termination |
|---|---|---|---|---|
| Cohort 1 | xx-xxxx | 0 (None) | 1 (Mild) | 1 (Mild) |
| Cohort 2 | | | | |
| Cohort 3 | | | | |
| Cohort 4 | | | | |

Created on: ddmmmyy hh:mm

L16.2.6.7 Listing of Application Site Reaction

| | | | | | Sign / Sy | mptom | | |
|---|---|---|---|---|---|---|---|---|
| Cohort | Patient<br>Number | Visit | Burning | Erosion | Edema | Pain | Itching | Dryness |
| Cohort 1 | XX-XXXX | 1 | 0 | 0 | 0 | 1 | 0 | 0 |
| | | 2 | 0 | 1 | 0 | 0 | 0 | 0 |
| | | 3 | 0 | 0 | 0 | 1 | 0 | 0 |
| Cohort 2 | | | | | | | | |
| Cohort 3 | | | | | | | | |
| Cohort 4 | | | | | | | | |

# L16.2.7 Listing of Adverse Events by Cohort

| Cohort | Patient<br>Number | Body System /<br>MedDRA Term /<br>AE Term | Treatment<br>Area | Start /End<br>Date | Severity | Relationship<br>to Study<br>Drug | Outcome | Action Taken/<br>Other Action<br>Taken | SAE? |
|---|---|---|---|---|---|---|---|---|---|
| Cohort 1 | xx-xxxx | Nervous system disorders /<br>Headache / | No | yyyy-mm-dd /<br>yyyy-mm-dd | Mild | Not Related | Recovered | Dose Not Changed/<br>None | No |
| | | Headache | | | | | | | |

Cohort 2

Cohort 3

Cohort 4

Related = Possible, Probable, Definite

Created on: ddmmmyy hh:mm

## L16.2.8.1 Listing of Positive Pregnancy Test Results

| Cohort | Patient<br>Number | Visit 1 | Visit 2 | Visit 3 |
|----------|-------------------|----------|----------|----------|
| Cohort 1 | xx-xxxx | Negative | Negative | Negative |
| Cohort 2 | | | | |
| Cohort 3 | | | | |
| Cohort 4 | | | | |

Created on: ddmmmyy hh:mm

## L16.2.8.2 Listing of Abnormal Vital Signs

| Cohort | Patient<br>Number | Age | Visit | Vital Sign | Normal Range | Result |
|---|---|---|---|---|---|---|
| Cohort 1 | xx-xxxx | xxx | 1 | Diastolic BP | xxx - xxx | XXX |
| | | | 2 3 | | | |
| Cohort 2<br>Cohort 3<br>Cohort 4 | | | | | | |

Created on: ddmmmyy hh:mm

L16.2.8.3 Listing of Abnormal Physical Examination Results

| Cohort | Patient<br>Number | Visit | System | Results |
|----------|-------------------|-------|--------|-----------------|
| Cohort 1 | xx-xxxx | 1 | HEENT | Abnormal (Scar) |
| | | 2 | | |
| | | 3 | | |
| Cohort 2 | | | | |
| Cohort 3 | | | | |
| Cohort 4 | | | | |

## L16.2.8.4 Listing of Clinical Hematology Laboratory Results

| Cohort | Patient<br>Number | Visit | Hematocrit (unit) | WBC (unit) | Platelets (unit) | Hemoglobin<br>( <i>unit</i> ) | etc. |
|---|---|---|---|---|---|---|---|
| Cohort 1 | XX-XXXX | 1 | xxx | XXX | XXX | XXX | XXX |
| | | 3 | xxx | xxx | XXX | xxx (Low) | XXX |

Cohort 2

Cohort 3

Cohort 4

Created on: ddmmmyy hh:mm

## L16.2.8.5 Listing of Clinical Chemistry Laboratory Results

| Cohort | Patient<br>Number | Visit | Alkaline<br>Phosphatase<br>( <i>unit</i> ) | Alnine<br>Transaminase<br>( <i>unit</i> ) | Aspartate<br>Transaminase<br>(unit) | Blood Urea<br>Nitrogen<br>( <i>unit</i> ) | etc. |
|---|---|---|---|---|---|---|---|
| Cohort 1 | xx-xxxx | 1 | XXX | XXX | xxx (High) | XXX | XXX |
| | | 3 | XXX | XXX | XXX | XXX | XXX |

Cohort 2

Cohort 3

Cohort 4

Created on: ddmmmyy hh:mm

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502a / 71615002

#### 10. APPENDICES

**APPENDIX A: Body Surface Area Calculation** 

#### **Total Body Surface Area Calculation**

To calculate the Total BSA the following procedure (Mosteller Formula<sup>13</sup>) should be followed.

Total Body Surface Area (BSA) in meters squared

$$m^2 = ((height (cm) x weight (kg)) / 3600)^{1/2}$$

It is preferable that the patient's height and weight be measured in cm and kg however if needed:

To convert inches (in) to centimeters (cm) the following conversion should be used

$$1 \text{ inch} = 2.54 \text{ cm}$$

To convert pounds (lbs) to kilograms (kg) the following conversion should be used

$$1 lb = 0.45 kg$$

The patient's height and weight should be reported to the nearest cm and nearest 0.5 kg. The BSA should be reported to the nearest second decimal place.

For example a patient who is 68 inches tall and weighs 180 lbs will have a reported BSA of:

#### **%BSA Affected**

To estimate the % BSA Affected, the Investigator should use the method of approximation:

The "Rule of Nines" provides a general estimation of total BSA for several anatomic areas (each arm = 9%, each leg = 18%, back = 18%, chest and abdomen = 18%, head =

# **Desoximetasone 0.15% Topical Spray**

Protocol / Study No. DSXS 1502a / 71615002

9%, groin = 1%). The Investigator may then visually estimate the proportion of the involved skin within each anatomic area and calculate the total percentage of BSA affected. In children, hips and legs are smaller and the head, neck and shoulders are larger, as a result, a modified "Rule of Nines" is used (see diagram below).

| Part | 1-4 year child<br>body<br>% of total | 5-9 year child<br>body<br>% of total | 10-14 year child<br>body<br>% of total | Adult body % of total |
|---|---|---|---|---|
| Arm | 9.5% | 9.5% | 9.5% | 9% |
| Head | 19% | 15% | 12% | 9% |
| Neck | 1970 | 1370 | 1% | 1% |
| Leg | 15% | 17% | 18% | 18% |
| Anterior trunk | 16% | 16% | 16% | 18% |
| Posterior trunk | 16% | 16% | 16% | 18% |



**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502a / 71615002

#### APPENDIX B: Eczema Area and Severity Index Score (EASI)

The EASI is a composite score based on the severity of four different signs of atopic dermatitis in four different areas of the body multiplied by the percent of that specific body area affected multiplied by a weighting factor.

Erythema

0 = Clear No evidence of erythema 1 = Mild Definite light red coloration 2 = Moderate Moderate redness, but not dark

3 = Severe Dark red coloration

Induration/papulation/edema

0 = Clear No evidence of any induration/papulation/edema

1 = Mild
2 = Moderate
3 = Severe

Barely perceptible elevation
Clearly perceptible elevation
Marked and extensive elevation

Lichenification

0 = Clear No evidence of lichenification

1 = Mild Slight thickening of skin discerible only by touch and with

skin markings minimally exaggerated

2 = Moderate Definite thickening of skin with skin marking exaggerated so

at they form a visible criss-cross or ridged pattern

3 = Severe Thickened skin with skin markings visibly portraying an

exaggerated criss-cross or ridged pattern

Excoriation

0 = Clear No evidence of excoriation

1 = Mild Scant evidence of excoriation with no signs of deepers skin

damage (absence of erosion or crusts)

2 = Moderate Several linear marks of skin with some showing evidence of

deeper skin injury (erosion, crust visible)

3 = Severe Many erosive or crusty lesions present

The patient will be required to rate the severity of their pruritis (itching/scratching/discomfort) over the previous 24 hours using the following scale:

**Pruritis** 

0 = None None

1 = Mild Occasional slight itching or scratching

2 = Moderate Constant or intermittent itching/scratching/discomfort which

is not disturbing sleep

## **Desoximetasone 0.15% Topical Spray**

Protocol / Study No. DSXS 1502a / 71615002

3 = Severe

Bothersome itching/scratching/discomfort which is disturbing sleep

Eczema, induration, excoriation and lichenification are part of the EASI score but pruritis is not.

#### **EASI Score**

The EASI score is calculated as follows:

Head/neck  $(E + I + X + L) \times Area \times 0.1$  (in children ages 0-7, x 0.2)

Upper Limbs (E+I+X+L) x Area x 0.2 Trunk (E+I+X+L) x Area x 0.3

Lower Limbs  $(E + I + X + L) \times Area \times 0.4$  (in children ages 0-7, x 0.3)

EASI SCORE = SUM OF ABOVE 4 REGIONS

E: Erythema,

I: Induration/papulation/edema

X: Excoriation

L: Lichenification

Severity is based on the Investigator's assessment of individual signs and symptoms 0 = none, 1 = mild, 2 = moderate, 3 = severe using the definitions above

The % of each body region affected is scored as the variable Area above in the EASI formula. For the 4 body regions (head/neck, upper limbs, trunk and lower limbs) if the:

```
Area = 0 if % affected is 0%

Area = 1 if % affected is 1 to 9%

Area = 2 if % affected is 10 to 29%

Area = 3 if % affected is 30 to 49%

Area = 4 if % affected is 50 to 69%

Area = 5 if % affected is 70 to 89%

Area = 6 if % affected is 90 to 100%
```

EASI Score can be presented to the nearest whole number (no decimals and all numbers should be rounded, 0.5 should be rounded up to the nearest whole number)

The minimum score would be 0 and the Maximum Score would be 72. To be eligible for participation in this study a patient must have an EASI of at least 15 at baseline.

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502a / 71615002

## **APPENDIX C: Investigator Global Assessment (IGA)**

To be eligible for inclusion in the study the IGA must be 3 or 4 at baseline. To be considered a Clinical Success the patient must score a 0, 1 at Visit 4.

| 0 | Clear | Minor, residual discoloration, no erythema or induration/papulation, no oozing/crusting |
|---|---|---|
| 1 | Almost Clear | Just perceptible erythema, with almost no induration/papulation and no oozing/crusting |
| 2 | Mild Disease | Definite pink erythema with mild induration/papulation and no oozing/crusting |
| 3 | Moderate<br>Disease | Red erythema with moderate induration/papulation and there may be some oozing/crusting |
| 4 | Severe<br>Disease | Dark/bright red erythema with severe induration/papulation with oozing/crusting |

**Desoximetasone 0.15% Topical Spray** 

Protocol / Study No. DSXS 1502a / 71615002

#### **APPENDIX D: Cortisol Response Test**

This cortisol release test is modified from the procedure of Wood et al as described in the Product Label for Cortrosyn<sup>TM</sup> (cosyntropin) for injection (Amphstar Pharmaceuticals, Inc.).

The procedure is as follows:

- 1. A single 5 ml blood sample should be taken as the basal sample.
- 2. 0.25 mg (a single vial) of Cortrosyn<sup>TM</sup> (cosyntropin) should be reconstituted with 1.0ml of 0.9% sodium chloride injection USP injected intramuscularly. In patients under 3 years of age, 0.125mg of Cortrosyn<sup>TM</sup> will be used.
- 3. 30 minutes after the IM injection a second 5 ml blood sample should be obtained. The resulting two serum samples (at least 1 ml of serum in each) should be processed and labeled according to the instructions provided and sent the same day to ACM Global Laboratory for analysis of basal and post stimulated serum cortisol concentration.

At Visit 1 and Visit 4 all patients will have a cortisol response test performed. The resulting blood sample should be sent to ACM Global Laboratory for immediate testing.

#### Visit 1 Test

The results of the cortisol response test must be obtained prior to study drug being dispensed at Visit 2. Only patients with normal baseline (Visit 1) cortisol and adrenal function (see criteria below) should be enrolled in the study.

#### Visit 4 Test

The test at the End of Study visit should not be performed if the patient dosed within 12 hours.

A patient will be considered to have normal basal cortisol level and adrenal function if they meet all three criteria listed below under Normal. Failure to meet any of these criteria is indicative of abnormal adrenal function or potential HPA axis suppression.

| | Cortisol Results | |
|---|---|---|
| | Normal | Abnormal |
| Basal (pre Cortrosyn <sup>TM</sup> injection) | ≥ 5 mcg/100ml | < 5 mcg/100ml |
| 30 minutes post<br>Cortrosyn <sup>TM</sup> | ≥ basal value + 7 | < basal value + 7 |
| Cortrosyn <sup>TM</sup> injection | > 18 mcg/100ml | ≤ 18 mcg/100ml |

HPA Axis suppression will be defined as a 30 minute post Cortrosyn<sup>TM</sup> injection level cortisol level of  $\leq$  18 mcg/100ml. As the study treatment period will be over, any patients with results of

## **Desoximetasone 0.15% Topical Spray**

Protocol / Study No. DSXS 1502a / 71615002

HPA axis suppression will be advised not to initiate any new steroid therapy, topical or otherwise, and to return to the site in 28 days at which time they will be assessed for HPA axis suppression.

Any patient presenting with symptoms of HPA axis suppression, such as nausea, headache, myalgia, fatigue or loose stool, will be referred to an endocrinologist. As an additional safety precaution, wristbands identifying the patient as someone suffering from adrenal suppression secondary to steroid withdrawal will be provided to alert medical personnel should any emergencies arise before adrenal function returns to normal.

If the results of the cortisol response test still show signs of HPA axis suppression 28 days after discontinuing therapy the patient will be asked to return in 28 days (56 days after discontinuing steroid therapy) for another follow-up test. If the patient is still showing signs of HPA axis suppression 56 days after discontinuing steroid therapy and presents with related symptoms, the patient will be referred to an endocrinologist.

If HPA axis suppression persists for 56 days after discontinuing steroid therapy, but the patient has no symptoms they will be asked to return in 28 days (84 days after discontinuing steroid therapy) for another follow-up test. If HPA axis suppression persists for 84 days after discontinuing steroid therapy patients will be referred to an endocrinologist regardless of symptoms.

Patients should not be subjected to Cortrosyn<sup>TM</sup> testing, or any other challenge to their adrenal response, any sooner than 4 weeks from their last Cortrosyn<sup>TM</sup> test.

Follow-Up Schedule for Patients showing signs of HPA Axis Suppression

| Days<br>after d/c | HPA Results | Symptoms | Patient Course |
|-------------------|-------------|-----------|-----------------------------|
| 28 | Normal | N/A | Study over |
| 28 | Abnormal | Yes | Refer to endocrinologist |
| 28 | Abnormal | No | Repeat test in 28 days |
| 56 | Normal | N/A | Study over |
| 56 | Abnormal | Yes | Refer to endocrinologist |
| 56 | Abnormal | No | Repeat test in 28 days |
| 84 | Normal | N/A | Study over |
| 84 | Abnormal | Yes or No | Refer to an endocrinologist |